CLINICAL TRIAL: NCT01605357
Title: A Randomized, Open Label Clinical Trial of Sustained Hypernatremia for the Prevention and Treatment of Cerebral Edema in Traumatic Brain Injury
Brief Title: Hypernatremia for the Prevention and Treatment of Cerebral Edema in Traumatic Brain Injury
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Never started.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Brian P. Walcott, Surgeon - Department of Neurosurgery, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MGH-HH5
Record Dates: First submitted 2012-05-22; First posted 2012-05-24 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-12

CONDITIONS: Traumatic Brain Injury; Subdural Hematoma; Cerebral Contusion; Head Injury; Cerebral Edema
Keywords: Brain Injuries; Hematoma, subdural; Decompressive Craniectomy; Saline solution, hypertonic; Hypernatremia; Intracranial hemorrhages; Head Injuries, closed; Intracranial pressure; Brain edema; Critical care; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Wounds and Injuries; Physiological Effects of Drugs; Pharmacologic Actions
MeSH Terms: conditions — Brain Injuries, Traumatic; Hematoma, Subdural; Brain Contusion; Craniocerebral Trauma; Brain Edema; Brain Injuries; Hypernatremia; Intracranial Hemorrhages; Head Injuries, Closed; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Wounds and Injuries | interventions — Standard of Care; Saline Solution, Hypertonic; Mannitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Care (Active Comparator): Patients will be managed to maintain a goal serum sodium of > 135 mmol/L , a well recognized value in the management of severe traumatic brain injury.
  Interventions: Drug: Standard of care (hypertonic saline and mannitol; serum sodium)
- Induced Hypernatremia (Experimental): Patients will be treated with induced, sustained hypernatremia for 5 days following injury by using hypertonic saline to target a goal serum sodium of 150-160 mmol/L
  Interventions: Drug: Induced, sustained hypernatremia using hypertonic saline

INTERVENTIONS:
Drug: Induced, sustained hypernatremia using hypertonic saline — Patients in the experimental arm will receive hypertonic saline to target a serum sodium goal of 150 - 160 mmol/L. All hypertonic saline will be administered intravenously.
  Loading phase: Upon enrollment 23.4 % hypertonic saline (volume 20 cc) will be administered via a central venous catheter. A continuous infusion of 3% hypertonic saline will be administered at a rate of 30 cc per hour and titrated every six hours to target a serum sodium goal of 150-160 mmol/L.
  Maintenance phase: Titrate serum sodium to 150-160 mmol/L using continuous 3% hypertonic saline infusion.
  Discontinuation phase: After 5 days of completed therapy, begin to wean 3% hypertonic saline rate by 10cc every 6 hours. Discontinue hypertonic saline infusion after infusing at a rate of 20cc an hour for 6 hours.
  Bolus dosing of hypertonic saline and mannitol are to be administered at the discretion of the provider to treat elevated intracranial pressure based on practice guidelines
  Arms: Induced Hypernatremia
Drug: Standard of care (hypertonic saline and mannitol; serum sodium) — Bolus dosing of hypertonic saline and mannitol are to be administered at the discretion of the provider to treat elevated intracranial pressure based on practice guidelines. Hyponatremia ( serum sodium < 135 mmol/L) is to be corrected at the discretion of the provider.
  Arms: Standard Care

SUMMARY:
Cerebral edema is seen heterogenous group of neurological disease states that mainly fall under the categories of metabolic, infectious, neoplasia, cerebrovascular, and traumatic brain injury disease states. Regardless of the driving force, cerebral edema is defined as the accumulation of fluid in the brain's intracellular and extracellular spaces. This occurs secondary to alterations in the complex interplay between four distinct fluid compartments within the cranium. In any human cranium; fluid is contained in the blood, the cerebrospinal fluid, interstitial fluid of the brain parenchyma, and the intracellular fluid of the neurons and glia. Fluid movement occurs normally between these compartments and depends on specific concentrations of solutes (such as sodium) and water. In brain-injured states, the normal regulation of this process is disturbed and cerebral edema can develop. Cerebral edema leads to increased intracranial pressure and mortality secondary to brain tissue compression, given the confines of the fixed-volume cranium. Additionally, secondary neuronal dysfunction or death can occur at the cellular level secondary to the disruption of ion gradients that control metabolism and function.

While studies utilizing bolus dosing of hyperosmolar therapy to target signs or symptoms of increased intracranial pressure secondary to cerebral edema are numerous, there is a paucity of studies relating to continuous infusion of hyperosmolar therapy for targeted sustained hypernatremia for the prevention and treatment of cerebral edema. The investigators hypothesize that induced, sustained hypernatremia following traumatic brain injury will decrease the rate of cerebral edema formation and improve patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 - 60 years old)
* Severe traumatic brain injury with intracranial pressure monitoring
* Initial GCS 5-8 (obtained free of the effects of neuromuscular blockade or sedatives)
* Clearly defined time of injury no more than 8 hours before administration of study drug
* Written consent obtained from legally authorized representative (LAR)
* Severe swelling prone injury patterns:

  1. Contusion - frontal or temporal (> 20 cc)
  2. Acute convexity subdural hematoma with any evidence of midline shift

Exclusion Criteria:

* Patients undergoing emergent (within 15 minutes) or urgent neurosurgery (within 4 hours) following emergency department arrival (bedside procedures, such as intracranial pressure monitor placement are excluded)
* Posterior fossa lesions
* Penetrating brain injury
* Spinal column instability and/or spinal cord injury with neurological deficit
* Pregnant
* Concomitant severe nonsurvivable injury
* Acute renal failure ; Chronic renal failure (serum creatinine of > 2.5 mg/dL, history of ongoing dialysis, glomerular filtration rate <30mL/min/1.73 m2); Severe pulmonary edema; Severe heart failure; Severe liver failure (AST, ALT, or bilirubin > 2 times normal)
* Known use of warfarin, clopidogrel, prasugrel, cilostazol, heparin, low molecular weight heparin, heparinoids, abciximab or similar antiplatelet agents
* Treatment with another investigational drug within the prior 30 days
* Systolic blood pressure < 90 mm HG not responsive to fluid resuscitation
* INR > 1.4
* Hospitalization for brain injury or neurological disease within previous 3 years
* Admission serum sodium < 135 mmol/L
* > 8 hours from the time of injury to admission
* Fix/dilated pupil suspected to be secondary to brainstem compression
* Duret (brainstem) hemorrhage indicating brainstem herniation
* PaO2 < 60 mmHg on admission (when blood gases are drawn as standard of care)
* Prisoner or other persons unable to make a true, voluntary and uncoerced decision whether or not to participate in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Objective | 72 hours ; 120 hours ; 30 days
  The primary efficacy objective of this study is to assess whether patients with severe TBI treated with sustained hypernatremia will show a decrease in neuroimaging defined edema compared to patients treated as the current standard of care.
Primary Safety Objective | Through 30 days
  The primary safety objective is to assess the safety and tolerability of sustained hypernatremia compared to the goal of avoiding hyponatremia in patients with severe traumatic brain injury. Safety will be assessed by a review of the incidence of mortality and adverse events, as well as by analysis of relevant laboratory data.

SECONDARY OUTCOMES:
Short term neurological outcome | 30 days
  The secondary outcome measure of this study will be assess whether patients with TBI treated with sustained hypernatremia will benefit patients in terms of short term neurological outcome - defined as need for tracheostomy during principal admission.
  Other secondary outcome measures will be need for delayed craniectomy and cumulative dosage of bolus dosing hyperosmolar therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Brian P Walcott, MD, Study Chair — Massachusetts General Hospital; Brian V Nahed, MD, Principal Investigator — Massachusetts General Hospital; Sameer A Sheth, MD PhD, Study Director — Massachusetts General Hospital